CLINICAL TRIAL: NCT04800926
Title: Xavier Electromyographic Wheelchair Control for Limited Mobility Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Central Florida (Other)
Responsible Party: Principal Investigator, Bjorn E. Oskarsson, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-002369
Record Dates: First submitted 2018-12-28; First posted 2021-03-16 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Xavier wheelchair controller (Experimental): Surface electromyography control of wheelchair
  Interventions: Device: Xavier wheelchair controller

INTERVENTIONS:
Device: Xavier wheelchair controller — Controlling a wheelchair using the Xavier surface EMG system

SUMMARY:
The purpose of this study is to assess the functional mobility and self-reported satisfaction with the Xavier electromyography hands-free wheelchair control system in comparison with a standard joystick.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosis by revised el Escorial criteria (definite, probable or probable laboratory supported)
* Age 18-89
* Limited mobility with use of motorized wheelchair at screening-time
* Impairment of hand function limiting the use of a standard joystick control
* Caregiver willing to assist with transfers into wheelchair and application of controllers
* Ability to attend study visits with a motorized wheelchair
* Ability to communicate and answer patient reported outcome measure questions

Exclusion Criteria:

* Cognitive impairment prohibiting safe independent mobility as defined by an ALS-Cognitive Behavioral Screen (ALS-CBS) score of <10 or the opinion of the investigator
* A sensory impairment prohibiting safe independent mobility in the opinion of the investigator
* Allergy to adhesives or electrode gels (required for EMG electrodes)
* Skin breakdown over the temporalis muscle that would predispose to further breakdown and/or infection with electrodes
* Severe loss of facial muscle functionality or control that would preclude EMG electrode efficacy
* Subjects who do not have the capacity to consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test (WST) | approximately 3 days
  Questionnaire

SECONDARY OUTCOMES:
Drive test | approximately 3 days
  Driving around cones in a controlled environment

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Oskarsson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Background] Manero AC, McLinden SL, Sparkman J, Oskarsson B. Evaluating surface EMG control of motorized wheelchairs for amyotrophic lateral sclerosis patients. J Neuroeng Rehabil. 2022 Aug 14;19(1):88. doi: 10.1186/s12984-022-01066-8. PMID 35965311
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials